CLINICAL TRIAL: NCT01153555
Title: Fractional Flow Reserve and Intravascular Ultrasound RelationShip STudy: The FIRST Study
Brief Title: Fractional Flow Reserve and Intravascular Ultrasound RelationShip STudy
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: FIRST
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intermediate coronary lesions: Diagnostic device: FFR
  Diagnostic device: IVUS RF
  At participating centers, FFR and IVUS are standard of care diagnostic procedures for patients with intermediate (40-80% angiographic stenosis by visual estimate). Both modalities were used regularly for such patients whether or not they are participants in this clinical study. In FIRST, the decision to perform percutaneous coronary intervention (PCI) was left to the discretion of the investigator, and was not dictated by the clinical protocol.

SUMMARY:
This is a multi-center, prospective registry of patients with intermediate coronary lesions defined as a stenosis of 40-80% by angiography. Approximately 300 patients will be enrolled into the study at sites in the United States and Europe. There will be no follow up beyond hospital discharge in this study. A sub-group of 30 patients will undergo Adenosine MRI. The investigators hypothesize that Intravascular Ultrasound Radiofrequency (IVUS RF) anatomical criteria, such as minimal luminal area, plaque burden and virtual histology plaque type, can predict physiological ischemia by Fractional Flow Reserve (FFR).

DETAILED DESCRIPTION:
Patients undergoing cardiac catheterization must meet clinical inclusion and exclusion criteria and sign an informed consent. At the time of catheterization the patients will be further analyzed for eligibility using angiographic inclusion and exclusion criteria. Patients who fulfilled the clinical and angiographic criteria will undergo further imaging evaluation using an IVUS RF catheter (Volcano Therapeutics) and FFR wire (Radi or Volcano). The decision for treatment of any lesion will be at the operator's discretion. For patients enrolled at Washington Hospital Center and do not undergo percutaneous coronary intervention, an assessment with non invasive perfusion adenosine MRI also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent to participate in the study.
* Clinical indication for coronary angiography for stable or unstable angina

Specific Angiographic Inclusion Criteria:

* Patients required to have an intermediate coronary lesion (stenosis 40-80% by visual estimate) in one or more native, major epicardial coronary artery with reference diameter ≥2.5mm (visual estimate)
* The vessel(s) with the intermediate lesion must have no flow limiting lesions and must be available for imaging and must be considered safe for imaging evaluation.

Exclusion Criteria:

* Patient has had a documented acute ST-segment elevation myocardial infarction within the past 24 hours
* Decompensated heart failure or hypotension requiring intubation, inotropes, intravenous diuretics or intraaortic balloon counterpulsation.
* Renal dysfunction (creatinine clearance < 60 mL/min/1.73m2)
* Pregnancy or breast-feeding
* Standard contra-indications to MRI for implanted ferro-magnetic devices - i.e.: pacemakers, defibrillator (AICD), and aneurysm clips
* Body weight > 400lbs
* Left ventricular hypertrophy >1.5cm by by echocardiogram
* History of bronchospasm or asthma
* ECG evidence of conduction defect, including 2nd or 3rd degree AVB
* Patient has a known hypersensitivity, allergy or contraindication to gadolinium-based contrast agents.
* Prior participation in this study or patient is currently enrolled in another investigational use device or drug study that has not reached its primary endpoint. If the patient is enrolled in another study that is not investigational, required visits for that trial must not interfere with the conduct of this trial.

Angiographic Exclusion Criteria:

* Unprotected left main lesion location.
* Ostial lesion
* Angiographic evidence of severe calcification or marked tortuosity of the target vessel that would preclude safe imaging
* Lesion is located within or distal to an arterial or saphenous vein graft.
* Angiographic presence of thrombus in the lesion or vessel studied.
* Lesion in a vessel with <2.5 mm reference diameter or with more than one lesion in the vessel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients required to have an intermediate coronary lesion (stenosis 40-80% by visual estimate) in one or more native, major epicardial coronary artery with reference diameter ≥2.5mm (visual estimate)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Correlation between (Minimum Luminal Area) MLA and FFR | Day of Procedure
  The correlation between MLA and FFR; and the threshold value for MLA corresponding to an FFR < 0.8.

SECONDARY OUTCOMES:
Correlation between FFR and IVUS and VH parameters | Day of Procedure
  Correlation between FFR and various IVUS measurements (MLA,area stenosis, lesion length, plaque burden) and VH parameters (plaque type and presence of a TCFA)
Association of FFR and Cut-off of MLA | Day of Procedure
  Assess the association between FFR <0.75 and 0.8 and determined cut-off of MLA with presence of a Thin Cap Fibro-Atheroma(TCFA) and/or plaque burden ≥70%
Identify risk score model | 1 year
  To identify a risk score model taking into account IVUS measurements (MLA, plaque burden, area stenosis, lesion length) and VH parameters (plaque type and presence of TCFA) associated with FFR < 0.8

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washingtoon Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Waksman R, Legutko J, Singh J, Orlando Q, Marso S, Schloss T, Tugaoen J, DeVries J, Palmer N, Haude M, Swymelar S, Torguson R. FIRST: Fractional Flow Reserve and Intravascular Ultrasound Relationship Study. J Am Coll Cardiol. 2013 Mar 5;61(9):917-23. doi: 10.1016/j.jacc.2012.12.012. Epub 2013 Jan 23. PMID 23352786